CLINICAL TRIAL: NCT03063047
Title: CSD1603: A Crossover Study to Evaluate the Exposure to "Tar" and Nicotine From 100s Menthol Cigarette Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Collaborators: Davita Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD1603
Record Dates: First submitted 2017-02-20; First posted 2017-02-24 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD21871AA, PD21872AA (Active Comparator): Subjects will use PD21871AA for 1 week and then PD21872AA for 1 week.
  Interventions: Other: PD21871AA; Other: PD21872AA
- PD21872AA, PD21871AA (Active Comparator): Subjects will use PD21872AA for 1 week and then PD21871AA for 1 week.
  Interventions: Other: PD21871AA; Other: PD21872AA

INTERVENTIONS:
Other: PD21871AA — A 100s size menthol cigarette.
Other: PD21872AA — A 100s size menthol cigarette.

SUMMARY:
This study will evaluate exposure to "tar" and nicotine from two menthol cigarette products and provide a basis for comparing mouth-level exposure when smokers smoke the two cigarette products. Mouth-level exposure is the measurement of substance trapped in the cigarette butt after smoking the cigarette.

Other purposes of this study are to:

* Compare the plasma cotinine, a byproduct of your body's processing of nicotine, levels found in users after smoking each of two different cigarettes.
* Find out the daily mouth-level exposure to cigarette "tar" and nicotine from smoking each of two different cigarettes in adult smokers.
* Determine if certain measures of nicotine dependence change based on the type of cigarette smoked
* To compare product liking and intent to use it again.

DETAILED DESCRIPTION:
The study will consist of one group of approximately 32 adult subjects randomly assigned to the order in which they will smoke two study menthol cigarette products (including one comparator product and one test product). Subjects will smoke each study product exclusively for approximately one week prior to a test visit, with a different product smoked each week over a two-week period. Cigarette butts will be collected the day prior to each test visit for determination of MLE "tar" and nicotine levels. Blood samples will be collected at each test visit for determination of plasma cotinine levels. Subjects will provide responses to questions during each test visit to assess their cigarette smoking and cigarette butt collection behavior during the preceding day.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, understand, and willing to sign an Informed Consent Form (ICF).
* Generally healthy males and females, 21 years of age or older, at Screening-Enrollment Visit.
* Self-reports smoking at least seven cigarettes per day and inhaling the smoke.
* Usual brand of cigarette is one of the brand styles specified.
* Smoked usual brand for ≥ 3 months.
* Agrees to exclusively smoke the study cigarettes and not smoke or use any other tobacco or nicotine-containing products during the course of the study.
* Able to read and comprehend English.
* Able to safely perform the required study procedures, as determined by the Investigator.

Exclusion Criteria:

* Self-reported history of heart disease, kidney disease, asthma or any other lung disease, diabetes, liver disease, hypertension, or hypercholesterolemia.
* At risk for heart disease, i.e., obesity (body mass index [BMI] ≥ 40 kg/m2), as determined by the Investigator.
* Females ≥ 35 years of age currently using systemic, estrogen-containing contraception, or hormone replacement therapy.
* Postponing a decision to quit smoking (defined as planning a quit attempt within 30 days of the Screening-Enrollment Visit) to participate in this study.
* Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (NRT) (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within 30 days prior to the Screening-Enrollment Visit.
* Females who test positive for pregnancy, are pregnant or breastfeeding, or plan to become pregnant during the course of the study.
* Determined by the Investigator to be inappropriate for the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
Mouth-level exposure (MLE) "tar" per cigarette and MLE nicotine per cigarette. | 2 weeks
  To compare the per cigarette MLE parameters (MLE "tar" per cigarette and MLE nicotine per cigarette) from smoking PD21871AA with those from smoking PD21872AA in adult smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Yoon, FNP-C, Principal Investigator — Davita Clinical Research
Locations (1):
- DaVita Clinical Research, Lakewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] St Charles FK, Kabbani AA, Borgerding MF. Estimating tar and nicotine exposure: human smoking versus machine generated smoke yields. Regul Toxicol Pharmacol. 2010 Feb;56(1):100-10. doi: 10.1016/j.yrtph.2009.08.011. Epub 2009 Aug 31. PMID 19723554
- [Background] Fagerstrom K. Determinants of tobacco use and renaming the FTND to the Fagerstrom Test for Cigarette Dependence. Nicotine Tob Res. 2012 Jan;14(1):75-8. doi: 10.1093/ntr/ntr137. Epub 2011 Oct 24. No abstract available. PMID 22025545
- [Background] Shepperd CJ, St Charles FK St, Lien M, Dixon M . Validation of methods for determining consumer smoked cigarette yields from cigarette filter analysis. Beitr Tabakforsch Int. 2006;22:176-184.